CLINICAL TRIAL: NCT01642719
Title: Chronic Moderate Sleep Restriction in Older Long Sleepers and Older Average Sleepers
Brief Title: Chronic Moderate Sleep Restriction in Older Adults
Acronym: MSSS
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Michael Irwin, MD, Director, Cousins Center for Psychoneuroimmunology; Cousins Professor,Department of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1R01HL095799-01A2 (NIH); 1R01HL095799-01A2 (NIH)
Record Dates: First submitted 2012-07-13; First posted 2012-07-17 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Sleep Disturbance; Aging
Keywords: Sleep disturbance; Aging; Sleep restriction; Health status; Glucose tolerance; Inflammation
MeSH Terms: conditions — Parasomnias; Inflammation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non-sleep restriction (Placebo Comparator): Participants will be asked to maintain fixed bedtimes, wake-times, times in bed, and napping, consistent with each person's average baseline
  Interventions: Behavioral: Non-sleep restriction
- Sleep restriction (Experimental): Participants will be asked to reduce their time in bed (TIB) by 60 min below their median baseline TIB, and to maintain this sleep restriction every night for 12 weeks. For example, if they spend 9 hr TIB during baseline, they will reduce their TIB to 8 hr.
  Interventions: Behavioral: Sleep restriction

INTERVENTIONS:
Behavioral: Sleep restriction — Participants will be asked to reduce their time in bed (TIB) by 60 min below their median baseline TIB, and to maintain this sleep restriction every night for 12 weeks.
  Arms: Sleep restriction
Behavioral: Non-sleep restriction — Participants will be asked to maintain fixed bedtimes, wake-times, times in bed, and napping, consistent with each person's average baseline.
  Arms: Non-sleep restriction

SUMMARY:
Higher rates of mortality have been found both in short sleepers (< 6 hr/night) and long sleepers (> 8 hr/night), but there has been little experimental investigation of the effects of chronic, moderate sleep loss in long or average sleepers. Some scientists argue that older adults might be particularly vulnerable to negative effects of sleep loss, whereas other scientists argue that many older adults spend too much time in bed, and that moderate reduction of time-in-bed could help increase the quality of their sleep, and could even promote health and longevity, particularly in long sleepers. At 4 sites across the US, we will conduct a large (200 people), randomized, controlled, 5- year study to examine whether a 1-hour reduction of time spent in bed for 12 weeks has negative or positive effects on multiple health-related outcomes, including inflammation, sleepiness, body weight, mood, glucose regulation, quality of life, incidence of illness, and incidence of automobile accidents in older long sleepers as compared to older average sleepers.

DETAILED DESCRIPTION:
Epidemiologic studies have consistently shown that self -reported sleep durations of <7 hr and >8 hr are associated with increased mortality and morbidity. The risks associated with short sleep are consistent with a vast experimental literature indicating detrimental effects of profound sleep restriction. However, there has been little study of chronic moderate sleep restriction, which is far more common, and thus more important from a public health standpoint. The risks associated with long sleep have scarcely been experimentally examined, though epidemiological data suggest sleep restriction might promote health/longevity in long sleepers. Older adults might be more vulnerable than young adults to negative effects of further sleep impairment, perhaps particularly via inflammatory mechanisms. Negative effects might be at least as evident in long sleepers as in average sleepers if long sleep reflects underlying morbidity, as many have posited. On the other hand, older adults might tolerate (or benefit) from moderate sleep restriction. Older adults often tend to spend excessive time in bed (TIB), particularly long sleepers, and extra TIB could contribute to age-related sleep fragmentation and morbidity, which could be ameliorated with modest TIB restriction. The aims of this study are: (1) to examine the ability of older long sleepers and older average sleepers to adhere to 60 min TIB restriction; and (2) to contrast effects of 12 weeks of 60 min TIB restriction on health-related measures in older long vs. average sleepers. One hundred older adults (ages 60-80 yr) who report sleeping 8-9 hr per night and 100 adults of the same age range who report sleeping 6-7.25 hr per night will be examined at 4 experimental sites over 5 years. Following a 2-week baseline, participants will be randomly assigned to one of two 12-week treatment groups. (1) A sleep restriction group (n=60 long sleepers and n=60 average sleepers) will be assigned to a fixed sleep- wake schedule, in which time in bed is reduced precisely 60 min below each participant's baseline time in bed (TIB). (2) A control group (n=40 long sleepers and n=40 average sleepers) will have no sleep restriction, but will also follow a fixed sleep schedule. Sleep will be assessed continuously with actigraphy and a daily diary. Questionnaires will be answered. Measures will include body weight, glucose tolerance, sleepiness, depression, quality of life, psychomotor vigilance, incidence of automobile accidents, incidence of illness, and multiple markers of inflammation. Physical exams during weeks 2 and 6 of the intervention and a study ombudsman will further monitor potential adverse effects. Follow-up assessments will be conducted for 12 months. The proposed clinical trial will provide the most comprehensive Phase 1 assessment of risks and benefits of chronic moderate TIB restriction ever conducted.

ELIGIBILITY:
Inclusion Criteria:

* 60-80 years of age
* Sleeping an average of 8-9 hr per night for long sleeper (or)
* Sleep an average of 6.0-7.25 hr per night for short sleepers
* Able to designate a study partner that can speak on their behalf throughout the course of the study.

Exclusion Criteria:

* Reported average sleep duration of < 8.0 hr or > 9.0 hr for longer sleepers
* Reported average sleep duration of < 6 hr or > 7.25 hr for the average sleepers
* Spending > 30 min time in bed in the morning and/or night outside of the major sleep period (e.g., watching tv)
* Expected change in usual sleep duration in the near future (e.g., change in work schedule)
* Reported average napping of > 2 naps/day or total nap duration of > 90 min/day;
* Recent shift-work (previous 2 months) or travel across multiple time zones (previous 4 weeks), or plans for performing shift-work or transmeridian travel during the study time period;
* Severe sleep apnea (apnea-hyponea index of greater or equal 15);
* Obesity (body mass index ≥35);
* High daytime sleepiness (Epworth Sleepiness Scale ≥ 10);
* Depression (Quick Inventory of Depressive Sympotomology > or equal to 16);
* Use of hypnotics or other drugs prescribed to promote sleep;
* Alcohol dependence or drug use;
* Any medical, neurologic, or psychiatric illness causing long sleep;
* Factors associated with significant changes in inflammation, including several medical disorders (e.g., rheumatoid arthritis), medications (e.g., steroids) and current smoking;
* Any health or mental condition that would contraindicate participation in the rigors of the study

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-07-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in adherence to sleep restriction from baseline | Daily for 12 weeks
  Evaluation of ability to adhere to a 60 min time-in-bed restriction over 12 weeks

SECONDARY OUTCOMES:
Change in sleepiness from baseline | Every week for 12 weeks
  Evaluation of sleepiness by weekly self-report for 12 weeks
Change in health functioning from baseline | Every 2 weeks for 12 weeks
  Evaluation of health functioning by self-report for 12 weeks
Change in sleep quality from baseline | Every month for 12 weeks
  Evaluation of sleep quality by self report every month for 12 weeks
Change in measures of cognitive performance from baseline | Every month for 12 weeks
  Evaluation of cognitive performance including standardized tasks to assess attention every month for 12 weeks
Change in physical activity from baseline | Every 8 weeks for 12 weeks
  Evaluation of physical activity by waist actigraphy and self-report every 8 weeks for 12 weeks
Markers of glucose metabolism | Baseline and at 12 weeks
  Evaluation of glucose metabolism by fasting glucose, glucose tolerance test, and hemoglobin A1C at baseline and again at 12 weeks
Change in depressive symptoms from baseline | Every 2 weeks for 12 weeks
  Evaluation of depressive symptoms by self-report every 2 weeks for 12 weeks
Markers of inflammation | Baseline and at 12 weeks
  Evaluation of cellular and genomic markers of inflammation at baseline and at 12 weeks
Change in fatigue from baseline | Every 2 weeks for 12 weeks
  Evaluation of fatigue by self-report every 2 weeks for 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Yougstedt, Ph.d., Principal Investigator — University of South Carolina; Richard Bootzin, Ph.D., Principal Investigator — University of Arizona; Michael Irwin, M.D., Principal Investigator — University of California, Los Angeles; Giardin Jean-Louis, Ph.D., Principal Investigator — State University of New York - Downstate Medical Center
Locations (4):
- United States (4):
  - University of Arizona, Tucson, Arizona
  - UCLA Cousins Center for Psychoneuroimmunology, Los Angeles, California
  - SUNY Downstate Medical Center, Brooklyn, New York
  - University of South Carolina, Columbia, South Carolina

REFERENCES:
- See also: UCLA Cousins Center for Psychoneuroimmunology — http://www.semel.ucla.edu/cousins